CLINICAL TRIAL: NCT07101718
Title: Outcomes and Risk Factors for Liver Transplantation Using Significant Fibrotic Grafts: a Retrospective Cohort Analysis of the US National Database
Brief Title: Outcomes and Risk Factors for Liver Transplantation Using Significant Fibrotic Grafts
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiao Xu, Professor, Zhejiang University
Other Study IDs: CT-2025-ZJU-OBS07
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Liver Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No fibrotic: Liver transplant recipient receiving no fibrotic liver grafts.
  Interventions: Other: No intervention
- Mild fibrotic: Liver transplant recipient receiving mild fibrotic liver grafts.
  Interventions: Other: No intervention
- Significant: Liver transplant recipient receiving significant fibrotic liver grafts.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This is a multi-center study to investigate the impact of fibrotic liver greafts in liver transplant recipient.

ELIGIBILITY:
Inclusion Criteria:

patients receiving liver transplantation during the period from March 2015 to March 2024

Exclusion Criteria:

1. recipients under 18 years old
2. re-transplantation cases
3. multiorgan transplant cases, reduced-size or split LT cases
4. lacking follow-up records or graft biopsy records

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A total of 25419 patients underwent liver transplant were studied.
Sampling Method: Probability Sample
Enrollment: 25419 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival rates | January 2015 to December 2024
  The overall survival of liver transplant recipients.

SECONDARY OUTCOMES:
Graft survival rates | January 2015 to December 2024
  The graft survival of liver transplant recipients.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University school of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No